CLINICAL TRIAL: NCT01608711
Title: An Open-Label Phase 2 Study of AGS-1C4D4 in Pancreatic Cancer Subjects Previously Treated in Protocol 2008002
Brief Title: A Study of AGS-1C4D4 in Pancreatic Cancer Subjects Previously Treated in Protocol 2008002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agensys, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGS-1C4D4-12-3
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Pancreatic Cancer; Carcinoma, Pancreatic Ductal; Pancreatic Disease
Keywords: Gemcitabine; ASP6182; AGS-1C4D4; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal; Pancreatic Diseases | interventions — MK-4721; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AGS-1C4D4 plus gemcitabine (Experimental): Subjects will receive a maintenance dose of AGS-1C4D4 every 3 weeks (Q3W) in addition to the gemcitabine administration.
  Interventions: Biological: AGS-1C4D4; Biological: gemcitabine

INTERVENTIONS:
Biological: AGS-1C4D4 — Intravenous Infusion
  Other Names: ASP6182
Biological: gemcitabine — Intravenous Infusion

SUMMARY:
The purpose of this study is to continue the safety and immunogenicity of AGS-1C4D4 administered in combination with gemcitabine in subjects previously treated in protocol 2008002.

DETAILED DESCRIPTION:
Subjects will receive a maintenance dose of AGS-1C4D4 every 3 weeks (Q3W) in addition to the gemcitabine administration. If subjects have grade 4 adverse events considered to be related to AGS-1C4D4 at anytime during the study, AGS-1C4D4 treatment will be discontinued for that subject.

Subjects will continue to have their tumor status assessed by computerized tomography (CT) and magnetic resonance (MRI) scans according to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) guidelines every eight weeks (Q8W). Subjects without evidence of disease progression will continue to receive AGS-1C4D4 and gemcitabine until intolerability, disease progression or consent withdrawal.

Subjects who discontinue AGS-1C4D4 for any reason will undergo an end of study visit 4 weeks after their last AGS-1C4D4 infusion.

ELIGIBILITY:
Inclusion Criteria:

* Subject has stable disease or better per Response Evaluation Criteria in Solid Tumors (RECIST) criteria v.1.1. in Protocol 2008002

Exclusion Criteria:

* More than 6 weeks (2 doses) has lapsed from the time of the last infusion in AGS-1C4D4 Protocol 2008002
* Use of the following prohibited medications / therapies:

  * Monoclonal antibody therapy, other than AGS-1C4D4
  * Chemotherapy, other than gemcitabine
  * Investigational therapy other than AGS-1C4D4
  * Erlotinib (Tarceva)
* Any clinical condition which would not allow safe conduct of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-08-07 (Actual); Primary Completion 2015-11-16 (Actual); Study Completion 2015-11-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 31 months
  Grade 3 and 4 adverse events, treatment-related adverse events, serious adverse events and adverse events requiring discontinuation of AGS-1C4D4
Incidence of anti-AGS-1C4D4 antibody formation | Every 8 weeks (up to 31 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Agensys, Inc.
Locations (2):
- Site US116, Madison, Wisconsin, United States
- Site CA00203, Toronto, Canada